CLINICAL TRIAL: NCT04523961
Title: Prospective, Randomized, Double-blinded, Split-face Study Comparing Efficacy of Lidocaine 2.5%/Prilocaine 2.5% Cream Under Occlusion, and Lidocaine 23% /Tetracaine 7% Ointment for Anesthesia Prior to 1927nm Fractional Laser Treatment
Brief Title: Comparative Study of Two Topical Anesthetics Prior to Fractional Nonablative Laser Treatment of the Face
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elika Hoss, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-002677
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia, Local; Photodamaged Skin; Topical and Infiltration Anesthetic Toxicity
MeSH Terms: interventions — Lidocaine; Tetracaine; Ointments; Salicylic Acid; Prilocaine; Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2.5 g of lidocaine 23% / tetracaine 7% ointment (Active Comparator): Patients undergoing 1927 nm fractional thulium fiber laser treatment of the face for photodamage as part of normal clinical care will have randomly assigned half of the face applied with 2.5 g of lidocaine 23% / tetracaine 7% ointment without occlusion for 60 minutes.
  Interventions: Drug: 2.5 g of lidocaine 23% / tetracaine 7% ointment without occlusion
- 7.5 g lidocaine 2.5%/ prilocaine 2.5% cream (Active Comparator): Patients undergoing 1927 nm fractional thulium fiber laser treatment of the face for photodamage as part of normal clinical care will have randomly assigned half of the face applied with 7.5 g lidocaine 2.5%/ prilocaine 2.5% cream with occlusion for 60 minutes.
  Interventions: Drug: 7.5 g lidocaine 2.5%/ prilocaine 2.5% cream with occlusion

INTERVENTIONS:
Drug: 2.5 g of lidocaine 23% / tetracaine 7% ointment without occlusion — Topical anesthetic used to numb the skin prior to laser procedures
  Other Names: 23/7 ointment
  Arms: 2.5 g of lidocaine 23% / tetracaine 7% ointment
Drug: 7.5 g lidocaine 2.5%/ prilocaine 2.5% cream with occlusion — Topical anesthetic used to numb the skin prior to laser procedures
  Other Names: EMLA Cream
  Arms: 7.5 g lidocaine 2.5%/ prilocaine 2.5% cream

SUMMARY:
The purpose of this study is to determine the efficacy of lidocaine 2.5%/prilocaine 2.5% cream versus lidocaine 23%/tetracaine 7% ointment for topical anesthesia prior to a nonablative laser procedure.

DETAILED DESCRIPTION:
Lidocaine 23% / tetracaine 7% ointment and lidocaine 2.5%/ prilocaine 2.5% cream are both topical anesthetics that are used commonly to locally anesthetize the skin prior to laser procedures. With the increased use of powerful lasers for medical and cosmetic purposes, adequate pain control is necessary. This study will compare the efficacy of lidocaine 23% / tetracaine 7% ointment and lidocaine 2.5%/ prilocaine 2.5% cream in reducing self-reported pain after laser treatment. It will also aim to determine the amount of redness, burning and itching a patient experiences with each cream, and if any symptoms of lidocaine toxicity are experienced.

Prior to the procedure, we will randomly assign half of the face to be applied with 2.5 g of lidocaine 23% / tetracaine 7% ointment without occlusion and the other half of the face with 7.5 g lidocaine 2.5%/ prilocaine 2.5% cream with occlusion. After 60 minutes we will remove the creams with soap and water. Next, the patient will be treated with a fractional thulium fiber laser with a fluence of 20 millijoules and treatment level of 7-11. Standard post procedure instructions will be given, and surveys on symptoms and pain will be completed by both patient and investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in general good health.18 years of age or older.
* Undergoing 1927nm fractional thulium laser treatment.
* Fitzpatrick skin type I-IV with at least mild photodamage of the face by physician discretion.
* Subject has completed an appropriately administered informed consent process which includes signing the institutional review board (IRB) approved consent form.
* Willingness to have facial exams and digital photos performed of the face.
* Female patients will be either of non-childbearing potential defined as:
* Having no uterus;
* No menses for at least 12 months; or
* (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:
* Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device;
* Intrauterine coil;
* Bilateral tubal ligation;
* Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom);
* Abstinence (if practicing abstinence must agree to use barrier method described above if becomes sexually active);
* Vasectomized partner (Must agree to use barrier method described above if becomes sexually active with non-vasectomized).

Exclusion Criteria:

* Presence of incompletely healed wound or active skin disease within in treatment area.
* Pregnant, planning pregnancy or breastfeeding during the course of the study.
* Individuals who have ablative laser within 6 months; non ablative lasers, facial peels, or dermabrasion within 1 month.
* Individuals with known allergies or sensitivities to any of the ingredients of any topical products being used in this study (a list of the products with active and excipients will be provided below).
* Subjects with any pre-existing medical or psychological condition which, in the opinion of the investigator, would put them at increased risk due to study treatment or participation.
* Subjects who are unable to comprehend the study consent document or provide full written consent.
* Subjects who have taken isotretinoin within 3 months or systemic corticosteroids within 1 month.
* Subjects with history of severe cardiovascular disease, kidney disease, liver disease, uncontrolled diabetes, uncontrolled seizures, immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Self-reported pain after laser treatment | After laser treatment, approximately 60 minutes
  Measure using a self-reported 11 point (0-10) visual analog scale (VAS) score with higher score indicated greater pain intensity

SECONDARY OUTCOMES:
Self-reported itching after laser treatment | After laser treatment, approximately 60 minutes
  Number of participants to report itching sensation after use of lidocaine 23% / tetracaine 7% ointment and lidocaine 2.5%/ prilocaine 2.5% cream
Self-reported burning after laser treatment | After laser treatment, approximately 60 minutes
  Number of participants to report burning sensation after use of lidocaine 23% / tetracaine 7% ointment and lidocaine 2.5%/ prilocaine 2.5% cream

CONTACTS AND LOCATIONS:
Overall Officials: Elika Hoss, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials